CLINICAL TRIAL: NCT04244110
Title: Diacare Project: Pilot for the Analysis of Usability in the Use of the Diacare Project for People With DM2 and Their Professionals
Brief Title: Pilot for the Analysis of Usability in the Use of the Diacare Platform for People With Type 2 DM and Their Professionals
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Fundació TicSalut (Other)
Responsible Party: Principal Investigator, Rosa Mª Flores, Principal Investigator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: DIACARE
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; self-management; mHealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate the usability, utility and feasibility of the Diacare platform and the ability of users to use the platform and receive valuable information from it to help address the management of type 2 diabetes outside the healthcare environment.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a chronic disease that increases the risk of patients suffering from heart disease, embolisms and microvascular complications such as blindness, kidney failure and peripheral neuropathies. In order to achieve an optimum level of independence in their self care, it is essential that type 2 DM patients take responsibility for the situation and be actively involved in the control of their health. Technology can solve some of the current challenges of chronic diseases such as type 2 DM, and in fact there are studies that suggest that chronic diseases can be more manageable with the support of mHealth. In this context, the Diacare platform has been designed with the idea of improving the self-management and self-care of patients with type 2 DM in a more personalized and individual way. The Diacare platform consists of an application, a fitbit wristband for activity monitoring and a web platform for professionals. This research project wants to evaluate the usability, utility and feasibility of the Diacare platform and the ability of users to use the platform and receive valuable information from it to help address the management of type 2 diabetes outside the healthcare environment. For this, a total of 35 patients and their respective health professionals will be recruited for the study and will use the DIACARE platform for 3 months. The results of this pilot will be collected through qualitative and quantitative data through the DIACARE platform and from questionnaires that will be administered to patients and professionals and will allow the evaluation of the technology developed.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with type 2 DM based on clinical criteria
* People who own a Smartphone and have competences in the use of technology

Exclusion Criteria:

* People that cannot go to the primary care center
* People with cognitive deterioration
* People with limitations in the practice of physical exercise
* People with a life expectancy lower than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The selected participants will belong to a primary care center based at Hospitalet de Llobregat, Barcelona (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Usability of the Diacare platform | 3 months
  System Usability Scale (SUS) is a self-administered questionnaire to evaluate the usability of the developed tool.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Flores, MD, Principal Investigator — Institut Català de la Salut
Locations (1):
- CAP Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No